CLINICAL TRIAL: NCT03118414
Title: Effects of Physical Exercise, Virtual Reality and Brain Exercise on Balance of the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Thwe Zar Chi Htut, Principal Investigator, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8.2.2016
Record Dates: First submitted 2017-03-31; First posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Elderly
Keywords: Balance; Cognition; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Physical Exercise Group (Experimental): Physical Exercise (PE) is an intervention that aim to improve balance and muscle strength of the elders. It composed of 3 steps; warming up exercise, core content of the exercise (strength and balance training) and cool down exercise program.
  Interventions: Other: Physical Exercise
- Virtual Reality (Experimental): Virtual Reality (VR) VR is an intervention that aim to improve balance of the elders. It stimulates the auditory and visual function and concentration of the participants throughout the training. It composed of 10 games that included weight shifting from side to side, stepping into different directions, trunk flexion, extension and side bending, movements of the upper and lower limbs, and trunk twisting in this study.
  Interventions: Other: Virtual Reality
- Brain Exercise (Experimental): Brain Exercise (BE) BE is an intervention that aim to stimulate the cognitive function of the elders.
  It stimulates the executive function, planning, concentration, visual memory and eye-hand co-ordination of the participants throughout the training
  Interventions: Other: Brain Exercise
- Control Group (No Intervention): No Intervention: Healthy control No intervention was given to this group of participants. The control group was reminded not to participate in any other exercise or intervention program except their routine daily activities.

INTERVENTIONS:
Other: Physical Exercise — Participants were trained by exercise program based on their initial muscle strength and balance condition.
  They received a 30-minute exercise for 3sessions per week for 8 weeks in this study.
  Arms: Physical Exercise Group
Other: Virtual Reality — Participants were trained with the guidance of VR system.The participants will be asked to choose 6 games from the list before each 30-minute session, and were asked to choose the games to include the upper limbs, lower limbs, and also for both strength and balance challenges instead of choosing the games that need to use only upper limbs or lower limbs, and only for strength or balance gain.
  They received a 30-minute exercise for 3sessions per week for 8 weeks in this study.
  Arms: Virtual Reality
Other: Brain Exercise — Brain Exercise (BE) BE stimulates the executive function, planning, concentration, visual memory and eye-hand co-ordination of the participants throughout the training.For the brain exercise, participants needed to play cognitive stimulating games; Chinese Checker, Janga and Memory Matched pair game; in the sitting position. The participants needed to paly 10 minutes for each gamed and total duration of all 3 games was about 30 minutes in each session for 3sessions per week for 8 weeks in this study.
  Arms: Brain Exercise

SUMMARY:
The objectives of this study were to 1) compare balance of the elderly by Berg Balance Scale (BBS) and Timed Up and Go Test (TUG) among physical exercise, virtual reality, brain exercise and control groups after intervention, 2) compare cognitive function of the elderly by using Timed Up and Go Cognitive (TUGC) and Montreal Cognitive Assessment (MoCA) among physical exercise, virtual reality, brain exercise and control groups after intervention, 3) compare muscle strength of elderly by 5 Times Sit-To-Stand Test (5TSTST) and Hand Grip Strength (HG) among physical exercise, virtual reality, brain exercise and control groups after intervention, 4) compare fear of falling by using Fall Efficacy Scale-International (FES-I) among physical exercise, virtual reality, brain exercise and control groups after intervention, 5)investigate the perspective of exercise among physical exercise, virtual reality, brain exercise and control groups after intervention.

DETAILED DESCRIPTION:
This study used healthy elderly participants with the age of 65-85 years. Eighty-four elderly participants were recruited by announcing the study information at the elderly homes. Sample size calculation was performed using G*Power software (G*Power version 3.1.9.2, University Kiel, Germany). To our knowledge, no study compare the effects of physical exercise, virtual reality and brain exercise on balance of the elders. Based on previous finding on the effects of virtual reality on balance of the elderly, a total of 84 participants were required at confidence level (α) of .05 and power (1-β) of 0.80. Participants who were interested in participation underwent a screening process using inclusion-exclusion criteria and receive brief information regarding the study. If they met all inclusion criteria, the consent process was performed. To ensure they understood the study, they were simply asked regarding the study (i.e. objectives, benefits, etc.) before signing the consent form.

After the participants provided a written informed consent, all participants filled out the information sheet and demographic data were collected. After that, age matching with range of ± 5 years and random allocation to different studies groups were done. Pretest assessment for balance by BBS and TUG, cognitive function by TUGC and MOCA, muscle strength by 5 TSTST and Hand Grip Strength (HG) and fear of falling by FES-I and perspective of exercise by questionnaires were done and recorded by blinded assessor. In this study, random allocation of the participants to different study groups; physical exercise group (PE), virtual reality group (VR), brain exercise group (BE) and control group; was done by the medical doctor and intervention was given the physical therapist from the study area which is the elderly home. All the assessments were done by the principal researcher. The assessor was blinded to reduce the bias which might come from the assessor's expectation.

After that, all the participants from intervention groups were explained and demonstrated about the respective interventions until they clearly understand about the intervention program before commencing the intervention program. The PE, VR and BE groups got their respective intervention for 30 minutes per sessions, 3 non-consecutive days per week for 8 weeks. The control group was reminded not to participate in any other exercise or intervention program except their routine daily activities for 8 weeks. Participants from PE group needed to do the 5-minute warm-up, 20-minute core content (upper and lower limb strengthening exercises and balance challenging exercises), and 5-minute cool down exercise programs. For the virtual reality group, the participants were reminded to play the game according to the program and try to get as high a score as possible they can. This intervention program included 10 games. The participants were asked to choose 6 games from the list before each 30-minute session, and were asked to choose the games to include the upper limbs, lower limbs, and also for both strength and balance challenges instead of choosing the games that need to use only upper limbs or lower limbs, and were just for strength and balance gain. For the brain exercise, participants needed to play cognitive stimulating games; Chinese Checker, Jenga and Memory Matched pair game; in the sitting position. The participants needed to paly 10 minutes for each game and total duration for all 3 games was about 30 minutes. After 8-week study period, post-test assessments were done to find out the effect of interventions.

The statistical analyses were performed by using SPSS for windows version 18.0, statistical software package. The value of p<0.05 was considered to indicate statistical significance. As the objective of this study was to find out the effects of PE, VR and BE on balance, cognitive function, muscle strength and fear of falling in the elderly. Two-way mixed ANOVA was used to test the variance differences among the four groups with post-hoc analysis as appropriately. Prior to utilization of statistical tests, descriptive statistics were performed and statistical assumptions were tested. Transformation will be performed if the data were not normally distributed. Appropriate statistical tests (parametric vs. non-parametric) were performed to determine the effects of different interventions in this study on balance, cognitive function, muscle strength and fear of falling in the elderly. Post-hoc power analysis was also performed.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-85 years
* MMSE score >23
* Able to do their activities of daily living by themselves (Berthal Index (BI) sore =100)
* No severe or unstable cardiopulmonary problem and are physically fit to perform the intervention programs by the medical notes and recommendation of the medical doctor.

Exclusion Criteria:

* Had lower limb injuries within 6 months or marked deformity at lower limbs
* Having severe or active arthritis
* Having psychological problems
* Who have been treated with lower extremity joint surgery, such as joint arthroplasty or joint fusion or amputation
* Having neurological problems such as stroke, Parkinsonism etc.,
* Having severe visual problem or the problem which could not be corrected by lens or glasses e.g. cataract.
* Having symptomatic vestibular impairment (such as dizziness or vertigo during movement) and severe hearing impairment which cannot be corrected by hearing aids.
* Having uncontrolled hypertension or diabetes.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Balance | 8 weeks
  Berg Balance Scale was used to measure functional balance. 14-item scale designed to measure balance of the older adult in a clinical setting.
  Description:
  Scoring: A five-point scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level.
  Total Score = 56 Interpretation: 41-56 = low fall risk 21-40 = medium fall risk 0 -20 = high fall risk

SECONDARY OUTCOMES:
Perceptive of Exercise | At the end of 8-week intervention
  Perspective of Exercise by Questionaries. The rating consisted of 6 scales; number 1 represents the least and number 6 represents the most satisfactory, beneficial or happy.
Cognition | 8 weeks
  Montreal Cognitive Assessment to assess cognitive function of the elders.
  Description:
  Total score=30 Interpretation: >26/30 = normal cognition
Lower Limb Muscle Strength | 8 weeks
  5 Times Sit To Stand Test to measure lower limb muscle strength. The participant to sit with the back against the back of the chair and with his/her arms crossed over the chest. Then, the participant was instructed to stand up and sit down as quickly and safely as he/she can without using the arms. Time taken (in seconds) to accomplished the task is recorded by stop watch. The shorter time reflect the better performance.
Fear of falling | 8 weeks
  Fall Efficacy Scale-International to assess fear of falling of the elderly16-item scale designed to measure fear of falling of the older adult Scoring: A four-point scale, ranging from 1-4. 1 = not at all concerned, 2 = somewhat concerned, 3 = fairly concerned, 4 = very concerned.' Total Score = 64 Interpretation: 16-19 = low concern 20-27 = moderate concern 28-64 = high concern
Mobility Balance | 8 weeks
  Timed up and Go test to assess the mobility balance. Get up from the chair and walk at a comfortable and safe pace to a line on the floor 3 meters away, turn, return to the chair and sit down again.
  Time taken (in seconds) to accomplished the task is recorded. The shorter time to accomplished reflect the better performance.
Cognitive Function (Dual Task) | 8 weeks
  Timed up and Go Cognitive to assess cognitive function of the elders. Get up from the chair and walk at a comfortable and safe pace to a line on the floor 3 meters away, turn, return to the chair and sit down again while counting backward by threes from a randomly selected number between 20 and 100. Time taken (in seconds) to accomplished the task is recorded by stop watch. The shorter time reflect the better performance.
General Muscle Strength | 8 weeks
  Hand grip strength to measure general muscle strength. The participant need to squeeze the dynamometer with the maximum effort and hold for 3 seconds without moving other parts of the body. The researcher read and noted down the strength of the hand grip in kilograms.

CONTACTS AND LOCATIONS:
Overall Officials: Thwe Zar Chi Htut, PhDcandidate, Principal Investigator — Mahidol University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller KL, Magel JR, Hayes JG. The effects of a home-based exercise program on balance confidence, balance performance, and gait in debilitated, ambulatory community-dwelling older adults: a pilot study. J Geriatr Phys Ther. 2010 Apr-Jun;33(2):85-91. PMID 20718388
- [Background] Lee S, Shin S. Effectiveness of virtual reality using video gaming technology in elderly adults with diabetes mellitus. Diabetes Technol Ther. 2013 Jun;15(6):489-96. doi: 10.1089/dia.2013.0050. Epub 2013 Apr 5. PMID 23560480
- [Background] Lee YM, Jang C, Bak IH, Yoon JS. Effects of Computer-assisted Cognitive Rehabilitation Training on the Cognition and Static Balance of the Elderly. J Phys Ther Sci. 2013 Nov;25(11):1475-7. doi: 10.1589/jpts.25.1475. Epub 2013 Dec 11. PMID 24396214